CLINICAL TRIAL: NCT06229223
Title: Improving Screening and Follow Up for Suicidal Ideation and Behaviors Among Latinx Youth in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00378575; R34MH129771 (NIH)
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PALOMA (Experimental): Parents/guardians of youth who have been referred to and agree to participate in the intervention by the child's primary care provider will participate in a 2-month program consisting of 5-7 phone sessions with a community health worker focusing on safety planning, information/education, program solving and self-care. Research participants will be asked to complete a survey via phone at the beginning of the program and another at the end of the program. The participants may also be asked to participate in an additional interview about the participants experience during the study.
  Interventions: Behavioral: PALOMA

INTERVENTIONS:
Behavioral: PALOMA — Partnering with Parents of Adolescent Latinos on Mental Health Assistance

SUMMARY:
The objective of this proposal is to develop and pilot a systems-level strategy in pediatric primary care to enhance identification and management of suicidal ideation and behavior in Latinx youth, particularly those in immigrant families with parents who have limited English proficiency (LEP). The investigators will focus on the use of trained community health workers (CHWs) to increase clinic capacity and quality of suicide risk screening and early intervention, with a focus on safety planning, parent psychoeducation and care coordination.

Specific aims are 1: To develop site-specific implementation protocols for the integration of CHWs into SIB screening and safety planning for Latinx youth and the youths families; 2: To pilot the implementation of the program in a six-month open trial in four pediatric primary care practices representing a range of usual practice settings; and 3: To engage a stakeholder network to explore barriers and facilitators, including costs and billing strategies, to implementation of this approach across a broad range of pediatric primary care settings.

Parents/guardians of youth who have been referred to and agree to participate in the intervention by the child's primary care provider will participate in a 2-month program consisting of 6-8 phone sessions with a community health worker focusing on safety planning, information/education, program solving and self-care. Research participants will be asked to complete a survey via phone at the beginning of the program and another at the end of the program. The participants may also be asked to participate in an additional interview about the study.

ELIGIBILITY:
Inclusion Criteria:

* Youth has history of suicidal ideation/behavior or non-suicidal self-harm and
* Youth identifies as Latino/Latinx/Hispanic/Latin American and
* Guardian(s) speaks Spanish

Exclusion Criteria:

* None

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants Screened | Monthly for 9 months
  Percent of patients 10-18 years old screened for depression and suicidal ideation and behavior at clinic level
Feasibility as assessed by percent of sessions completed | Monthly for 9 months
  Percent of eligible patients receiving a CHW session
Quality as assessed by percent of CHW visits | Monthly for 9 months
  Percent of CHW visits that include delivery of one or more intervention components
Engagement as assessed by number of follow-up visits | Monthly for 9 months
  number of follow-up mental health visits with PCP or specialty provider among youth identified as having suicidal ideation or behavior.

SECONDARY OUTCOMES:
Family Functioning as assessed by the SCORE-15 Index of Family Functioning and Change (SCORE-15) | Baseline and 3 months
  SCORE-15 Index of Family Functioning and Change: Score range 5-15, higher total means worse functioning.
Parent Self Efficacy as assessed by Brief Parenting Self Efficacy Scale (BPSES) Questionnaire | Baseline and 3 months
  Brief Parenting Self Efficacy Scale (BPSES) Questionnaire: Total score ranges from 5 to 25, higher scores indicate higher levels of parental self-efficacy.
Depression as assessed by the Patient Health Questionnaire - Adolescent (PHQ-A) | Baseline and 3 months
  Patient Health Questionnaire - Adolescent (PHQ-A): Each item on the PHQ-A is scored as follows: Not at all = 0 Several Days = 1 More than half the days = 2 Nearly every day = 3. A weighted score of 5 or more means a positive screen for depressive symptoms. A weighted score of 0-4 means a negative screen for depressive symptoms.
Suicidal Ideation and Behavior as assessed by the Ask Suicide-Screening Questionnaire (ASQ) | Baseline and 3 months
  Ask Suicide-Screening Questionnaire (ASQ): 4 Yes or No Questions. "Yes" to questions 1 through 4, or refuses to answer is considered a positive screen. "Yes" to question 5 = acute positive screen (imminent risk identified); "No" to question 5 = non-acute positive screen.
Parental Self-Efficacy to Support Teens During a Suicidal Crisis survey | Baseline and 3 months
  9 items. Answer choices ranged from 0 (not at all confident) to 10 (completely confident), with an anchor of 5 (somewhat confident); score range 0-90; higher score higher confidence.
Parent expectations of adolescents' risk survey | Baseline and 3 months
  3 items. Answer choices ranged from 0 (not at all confident) to 10 (completely confident), with an anchor of 5 (somewhat confident). Score range 0-30; higher score higher confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Polk, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- BMS at Yard 56, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available while safeguarding the privacy of participants, & protecting confidential & proprietary data. Investigators will have access to results free from personal identifiers & PHI. Investigators will fill out a request form that specifies the purpose of the request, the data requested & the qualifications of the requestor. Final research data will include recorded factual material necessary to document & support research findings, including final data sets (w/ identifiers redacted), data collection protocols data, & database documentation. Users must agree to the conditions of use governing access to the publicly released data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, restrictions on use for commercial purposes, & proper acknowledgement of the data resource.